CLINICAL TRIAL: NCT07365982
Title: THE EFFECT OF PSYCHOEDUCATION-BASED MOTIVATIONAL INTERVIEWING ON KNOWLEDGE ABOUT SCHIZOPHRENIA AND HOPE LEVELS IN PATIENTS DIAGNOSED WITH SCHIZOPHRENIA
Brief Title: Effect of Psychoeducation -Based Motivational Interviewing on Knowledge and Hope in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Büşra Taşkıner (Other)
Responsible Party: Sponsor-Investigator, Büşra Taşkıner, Principal Investigator ,Graduate Student in Psychiatric Nursing, Okan University
Organization: Okan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OKAN-ETIK-2025-K8
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Psychoeducation; Motivational Interviewing; Knowledge Level; Hope
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either an intervention group or a control group and followed in parallel throughout the study period.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was blinded to group allocation during the pre-test, post-test, and follow-up assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation-Based Motivational Interviewing (Experimental): Participants received a psychoeducation-based motivational interviewing program consisting of one preparatory session followed by five main sessions, in addition to routine community mental health services.
  Interventions: Behavioral: Psychoeducation-Based Motivational Interviewing
- Control Group - Routine Community Mental Health Services (No Intervention): Participants received routine community mental health center services only, without any additional psychosocial or motivational interviewing intervention.

INTERVENTIONS:
Behavioral: Psychoeducation-Based Motivational Interviewing — A structured psychoeducation-based motivational interviewing program delivered in weekly sessions lasting approximately 60-90 minutes, consisting of one preparatory session followed by five main sessions.
  Arms: Psychoeducation-Based Motivational Interviewing

SUMMARY:
This study aimed to examine the effect of a psychoeducation-based motivational interviewing intervention on schizophrenia-related knowledge and hope levels among patients diagnosed with schizophrenia. The study employed a randomized controlled experimental design with pre-test, post-test, and one-month follow-up measurements. Participants were recruited from a community mental health center and assigned to an intervention group or a control group. The intervention group participated in a structured psychoeducation-based motivational interviewing program consisting of one preparatory session followed by five main sessions, while the control group continued to receive routine community mental health services. Knowledge about schizophrenia and hope levels were assessed using validated measurement tools.

DETAILED DESCRIPTION:
The present study aimed to examine the effect of a psychoeducation-based motivational interviewing intervention on schizophrenia-related knowledge and hope levels among patients diagnosed with schizophrenia. The study was conducted using a randomized controlled experimental design with pre-test, post-test, and one-month follow-up measurements.

A total of 44 patients diagnosed with schizophrenia were included in the study, with 21 participants assigned to the intervention group and 23 to the control group. The study was carried out with individuals followed at a community mental health center between January and June 2025.

Participants in the intervention group received a structured psychoeducation-based motivational interviewing program consisting of one preparatory session followed by five main sessions. The sessions were conducted at least once per week, and each session lasted approximately 60 to 90 minutes. Throughout the study period, the control group continued to receive routine community mental health services.

Data were collected using a Demographic Information Form, the Schizophrenia Knowledge Level Scale, and the Schizophrenia Hope Scale. Changes in knowledge and hope levels were evaluated across measurement points.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the study and provided informed consent
* Aged between 18 and 65 years
* Literate
* Diagnosed with schizophrenia according to DSM-5 diagnostic criteria
* In remission phase (not in an acute exacerbation period)

Exclusion Criteria:

* Presence of severe intellectual disability as documented in hospital records
* Diagnosis of dementia and/or other organic mental disorders
* Currently in an acute exacerbation phase
* Discontinuation of intervention sessions or failure to complete assessment forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Schizophrenia Knowledge Level | Baseline (pre-test) prior to the intervention, immediately after completion of the final intervention session (post-test), and 1 month after completion of the intervention (follow-up assessment).
  Change in schizophrenia-related knowledge level assessed using the Schizophrenia Knowledge Level Scale. The scale consists of multiple-choice items assessing knowledge about schizophrenia, with total scores ranging from 0 to 25. Higher scores indicate greater knowledge about schizophrenia.

SECONDARY OUTCOMES:
Schizophrenia Hope Level | Baseline (pre-test) prior to the intervention, immediately after completion of the final intervention session (post-test), and 1 month after completion of the intervention (follow-up assessment).
  Change in hope level assessed using the Schizophrenia Hope Scale. The scale is a Likert-type measure with total scores ranging from 0 to 18. Higher scores indicate higher levels of hope.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Aycanoğlu, Assoc. Prof. Dr., Principal Investigator — Okan University
Locations (1):
- Zeytinburnu Community Mental Health Center (TRSM), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as the study is conducted as part of a master's thesis and the data are collected solely for academic purposes. All data are kept confidential in accordance with ethical approval and institutional regulations.